CLINICAL TRIAL: NCT06180772
Title: FIT FIRST FOR ALL - The Dose-Response Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Southern Denmark (Other)
Collaborators: Novo Nordisk A/S (Industry); National Olympic Committee and Sports Confederation of Denmark (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: USouthernDenmark-FIT FIRST
Record Dates: First submitted 2022-12-12; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Primary Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Continue normal activities
- 3/wk (Experimental): Use FIT FIRST 3 times pr. week
  Interventions: Behavioral: FIT FIRST
- 1.5/wk (Experimental): Use FIT FIRST 1.5 times pr. week
  Interventions: Behavioral: FIT FIRST

INTERVENTIONS:
Behavioral: FIT FIRST — High intensity sports drills and games
  Arms: 1.5/wk; 3/wk

SUMMARY:
In the present study, FIT FIRST 10 will run over 20 weeks, with cardiometabolic fitness as the primary outcome and project acceptability as the co-primary outcome. In this study the investigators will be testing the dose-response of the FIT FIRST concept by having two experimental groups. This will be a cluster RCT with a 1:1:1 recruitment of control schools, intervention schools with 3 weekly 40-min FIT FIRST 10 lessons, and intervention schools with 1.5 weekly 40-min session. There will be recruited a total of 1000 children, with 500 8-9-year-olds from 2nd and 3rd grade in each group from a minimum of 40 classes from 16 schools. There will be subgroup analyses of children with low socioeconomic status and ethnic minority background. Intervention effects will be tested as on health profile, cardiometabolic and musculoskeletal fitness, motivation for physical activity, acceptability of the programme for stakeholders as well as the implementation potential. The study will be running in Q1 and Q2 in 2023.

It is hypothesized that the FIT FIRST 10 concept will improve the well-being, increase sports club participation as well as increase fitness and health levels among 8-9-year-old children with low fitness, low socioeconomic and/or ethnic minority background. However, it is also hypothesized that the effects on well-being and fitness levels caused by the intervention may be most significant among ethnic minority children not enrolled in sports clubs.

DETAILED DESCRIPTION:
Background Physical activity (PA) is an important part of a healthy lifestyle for children and youth, as it improves physical fitness, motor competences and well-being, and reduces the risk of developing overweight and lifestyle diseases later in life. Current recommendations from the Danish Health Authorities are that young people should participate in at least 60 min of moderate-to-vigorous physical activity (MVPA) per day, of which at least 3 times 30 min per week should involve vigorous physical activity (VPA).

As children's total amount of daily PA is a product of their activities in and outside of school, it can be of value to look for synergetic effects that can be achieved by having developed abilities and motivation for activities in school that can be used in leisure time sports clubs.

Based on the beforementioned knowledge, investigators have developed the FIT FIRST programme. FIT FIRST was originally an acronym for a 40-week intervention study for 8-9-year-olds: Frequent Intense Training through Football, Interval Running and Circuit Strength Training. This study showed that 3x40 min per week of FIT FIRST ball game and circuit strength training activities was very effective in improving fat percentage, blood pressure, muscle strength, postural balance and bone mineralization. In 2018, the FIT FIRST 10 concept was developed for 6-9-year-olds that covered 10 sports using the same principles.

In the present study, FIT FIRST 10 will run over 20 weeks with cardiometabolic and musculoskeletal fitness as the primary outcomes and project acceptability as co-primary outcomes. In this study the investigators will be testing the dose-response of the FIT FIRST 10 concept by having two experimental groups. This will be a cluster RCT with a 1:1:1 recruitment of control schools, intervention schools with 3 weekly 40-min FIT FIRST 10 lessons, and intervention schools with 1.5 weekly 40-min session. There will be recruited a total of 2400 children, with 800 8-9-year-olds from 2nd and 3rd grade in each group from approximately 60 classes from 24 schools. There will be subgroup analyses of children with low socioeconomic status and ethnic minority background.

Intervention effects will be tested as in Study I on health profile, cardiometabolic and muscular fitness, motivation for physical activity, acceptability of the programme for stakeholders, and implementation potential. The study will be running in Q1 and Q2 in 2023.

Measures:

Fitness levels and health profile:

Yo-Yo IR1 Children's test (total distance in meters) will be used to evaluate cardiometabolic fitness. For muscular fitness, the standing long jump test (in meters), the handgrip strength test (in kilograms), the arrowhead agility-test (in seconds) and the stork balance stand test (in seconds) will be used.

To evaluate the effects on health, measurements of resting heart rate (beats per minute) and blood pressure (millimeters of mercury) will be recorded.

Also, the participants' body composition and height will be measured using Tanita scales and InBody 230 Bioimpedance. The measurements of the participants' body composition includes measures of their body mass (in kilograms), skeletal muscle mass (in kilograms) and fat percentage. To investigate the prevalence of overweight and obesity, BMI z-scores (kg/m^2) will be calculated by using the participants' relative weight adjusted for child age and sex.

Well-being, body image, self-worth and quality of life:

KIDSCREEN 27, which is a validated questionnaire measuring physical well-being, mental well-being, social well-being and school well-being in the school environment will be used. Children's body perception and satisfaction will be measured using the Children's Body Image Scale, a pictorial scale developed for 7-11 year old children. Furthermore, the short form of the Physical Self-Inventory (PSI-S) will be used to evaluate overall selfworth (i.e., perceptions of one's physical self) and specific sub-components (physical appearance, strength, physical condition and sport competence).

Evaluation of physical activity and sport club participation:

A questionnaire will provide information in terms of types of activities undertaken outside school.

Process evaluation:

The RE-AIM framework will be used to ensure a holistic assessment of intervention and implementation outcomes. A mixed-method approach, including document analysis, participant observations, objective measurements, survey instruments and interviews will be applied. The RE-AIM framework has been used extensively to assess school-based PA interventions and to guide process evaluations. The RE-AIM have been in several studies. The framework constitutes five key elements, i.e. Reach, Effectiveness, Adoption, Implementation and Maintenance.

Also, the ecological model of implementation, by Durlak and Dupree will be used.

ELIGIBILITY:
Inclusion Criteria:

* part of enrolled classes

Exclusion Criteria:

* none

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2400 (Estimated)
Dates: Start 2022-12-10 (Actual); Primary Completion 2024-12-24 (Estimated); Study Completion 2024-12-24 (Estimated)

PRIMARY OUTCOMES:
Cardiometabolic fitness as assessed by the achieved distance in the Yo-Yo IR1 Children's test | Change from baseline to week 20
  Cardiometabolic fitness profile will be evaluated by using the Yo-Yo IR1 Children's test measured as the total distance in meters as an indicator for the participants' ability to perform intermittent exercise and their cardiometabolic fitness. The longer the distance, the better the cardiometabolic fitness of the participants.
Project acceptability as assessed by observations and teachers questionnaires | Change from baseline to week 20
  Observations will describe the acceptability and specific teacher questionnaires will be applied to evaluate the acceptability of the project.

SECONDARY OUTCOMES:
Muscle strength of the lower body as assessed by the standing long jump performance | Change from baseline to week 20
  For muscular strength of the lower body, the standing long jump test will be used. The outcome will be the jumped distance measured in meters. The standing long jump test is applied to asses the lower body strength of the participants and the higher the score, the better the performance. The participants have to attempts.
Well-being as assessed by the questionnaires KIDSCREEN 27 | Change from baseline to week 20
  To evaluate the participants' well-being, - KIDSCREEN 27
Fat percentage based on bioimpedance. | Change from baseline to week 20
  To evaluate the effects on Fat percentage, bioimpendance will be used
Postural balance as assessed by the stork balance stand test | Change from baseline to week 20
  The stork balance stand test, measured three times on each leg, will be used to evaluate the participants' ability to maintain a state of balance in a static position. The outcome is measured in seconds and a higher score indicates a better outcome.
Agility as assessed by the arrowhead agility-test | Change from baseline to week 20
  The arrowhead-agility test is applied to assess the agility of the participants, their body control and change of direction. In this test, the participants have to attempts and will be running to the right side in both attempts. The outcome is measured in seconds. A lower score indicates a better outcome.
General strength as assessed by the handgrip strength test | Change from baseline to week 20
  The handgrip strength test is used to asses the participants' general strength level, measured in kilograms. A higher score indicates a better general strength. The participants have to attempts and use their dominant arm.
Health profile as assessed by resting heart rate | Change from baseline to week 20
  To evaluate the effects on health, measurements of resting heart rate (beats per minute).
Muscle mass | Change from baseline to week 20
  To evaluate the effects on Muscle mass, bioimpendance will be used.
systolic and diastolic blood pressure | Change from baseline to week 20
  systolic as well as diastolic blood pressure (millimeters of mercury) will be recorded three times with an automatic BP-monitor (M6 HEM-7322U-E; Omron, Hoofddorp, The Netherlands).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Krustrup, Principal Investigator — Syddansk Universitet - Sport og Sundhed (IOB)
Locations (1):
- University of Southern Denmark, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No